CLINICAL TRIAL: NCT02912741
Title: Double Blinded Randomized Clinical Trial for Evaluation of Resin Modified Glass Ionomer Cement Versus Resin Infiltration in Treating White Spot Lesions
Brief Title: One Year Clinical Evaluation of White Spot Lesions Treated With Newly Introduced Resin Modified Glass Ionomer in Comparison to Resin Infiltration in Anterior Teeth Split Mouth Technique
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Mostafa Rohym, Specialist in Air-Force Specialized Hospital, New Cairo, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-209
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: White Spot Lesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vanish xt Extended Contact Varnish (Experimental): Vanish xt Extended Contact Varnish is a resin modified glass ionomer cement and fluoride varnish used to treat white spot lesions to be more resistant to early caries progression.
  Interventions: Drug: Vanish xt Extended Contact Varnish
- Resin infiltration (Active Comparator): Resin infiltration is a low viscous resin infiltrates into small pores of white spot lesions to block entrance of bacteria into dentinal tubules of the tooth and more resistant to early caries progression.
  Interventions: Drug: resin infiltration

INTERVENTIONS:
Drug: Vanish xt Extended Contact Varnish — resin modified glass- ionomer cement varnish applied as a thin layer coating and cured
  Other Names: Clinpro xt
  Arms: Vanish xt Extended Contact Varnish
Drug: resin infiltration — low viscous light cure resin applied in layers and cured
  Other Names: ICON
  Arms: Resin infiltration

SUMMARY:
The aim of this study is to evaluate the addition of new technology of resin modified glass-ionomer in comparison to resin infiltration in treating post-orthodontic white spot lesions; both applies into the same patient's mouth; to reveal which material will have more clinical satisfactory performance inside the oral cavity and to overcome the high expensive cost in treating such clinical cases

DETAILED DESCRIPTION:
Roles and responsibilities:

* Shaimaa Mohammed (SH.M.): Operator and author.Specialist in Air-Force Specialized Hospital.
* Mohamed Riad (M.R.): Main supervisor, data monitoring and auditing, Professor, Conservative Dentistry Department,Cairo University.
* Asma Harhash(A.H.):Co-supervisor, outcome assessor and data collection, Associate Professor, Russian University.
* Omnia Magdy Moustafa (O.M.): Baseline data collection, recruitment, sequence generation, allocation concealment, patient retention and taking participants consents: Assistant lecturer, Conservative Dentistry Department , Faculty of Oral and Dental Medicine Cairo University.
* Ghada Ahmed (G.A.): Data entry and auditing; Assistant lecturer, Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Russian University.

Intervention:

A- Preoperative clinical assessment:

1. Explain patient need toward aesthetic needs
2. Digital photos for white spot lesions
3. Recording number of white spot lesions and site. (SH.M.) will apply both materials at the same patient mouth (Split mouth technique) according to the manufacturer's instructions.

   * Intervention: resin modified glass ionomer cement varnish: Vanish™ xt Extended Contact Varnish (3M ESPE Dental)
   * Comparator: resin infiltration (Dental Milestones Guaranteed, Germany).

(A.H) and (SH.M) will assess the outcome measures through the follow up time: immediately after,1 day, 1 week,1 month,3 months, 6 months, 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Post-Orthodontic patients included in this clinical trial toll age of 35 years.
2. Patients with good general health.
3. Patients who will agree to the consent and will commit to follow-up period.
4. Fully erupted anterior teeth with no cavitated lesions.
5. At least one spot lesion on each side in the same jaw

Exclusion Criteria:

1. Patients with any systemic disease that may affect normal healing.
2. Patient with bad oral hygiene.
3. Tetracycline or fluorsis staining.
4. Patients who could/would not participate in all times of follow-up.
5. Untreated periodontal disease was not allowed.
6. Active caries or defective Restorations in 6 anterior teeth.
7. Bleaching history
8. Patients participating in more than 1 dental study.
9. Patient received fluoride varnish during orthodontic treatment.

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in Patient satisfaction | immediately, 1 day, 1week,1 month,3 month,6 month and1 year
  using visual analogue scale ruler (0-100 mm) 0 refer to not satisfied at all,100 refer to total satisfied

SECONDARY OUTCOMES:
Change in color change | immediately, 1 day, 1week,1 month,3 month,6 month and1 year
  using vita easy shade device

OTHER OUTCOMES:
Change in caries lesion state | immediately, 1 day, 1week,1 month,3 month,6 month and1 year
  Diagnodent device

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkhadem, PhD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided